CLINICAL TRIAL: NCT00479882
Title: A Multicenter, Randomized, Double-Blind, "Crossover" Design Study to Evaluate the Lipid-Altering Efficacy and Safety of MK-0524B Combination Tablet Compared to MK-0524A + Simvastatin Coadministration in Patients With Primary Hypercholesterolemia and Mixed Dyslipidemia
Brief Title: MK-0524B Lipid Study (MK-0524B-063)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0524B-063; MK-0524B-063 (Other: Merck Study Number); 2007_504
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Results first posted 2016-04-01 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-01

CONDITIONS: Primary Hypercholesterolemia; Mixed Dyslipidemia
MeSH Terms: interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1: MK-0524B 1.8g/20mg→MK-0524A 2g+Simvastatin 20mg (Experimental): After a 2-week placebo run-in, participants will receive MK-0524B (0.9 g/simvastatin 10 mg) for 4 weeks, then MK-0524B 1.8g /20 mg combination tablet for 8 weeks. Participant is then co-administered MK-0524A 2 g + simvastatin 20 mg for 8 weeks.
  Interventions: Drug: Comparator: simvastatin; Drug: MK-0524A; Drug: Placebo; Drug: MK-0524B
- Sequence 2: MK-0524A 2g+Simvastatin 20mg →MK-0524B 1.8g/20mg (Experimental): After a 2-week placebo run-in, participants will be co-administered MK-0524A 1g + simvastatin 10 mg for 4 weeks, then co-administered MK-0524A 2g +simvastatin 20 mg for 8 weeks. Participant then receives MK-0524B 1.8 g/20 mg combination tablet for 8 weeks.
  Interventions: Drug: Comparator: simvastatin; Drug: MK-0524A; Drug: Placebo; Drug: MK-0524B
- Sequence 3: MK-0524B 1.8g/40mg→MK-0524A 2g+Simvastatin 40mg (Experimental): After a 2-week placebo run-in, participants will receive MK-0524B 0.9g/40 mg combination tablet for 4 weeks, then MK-0524B 1.8g /40 mg combination tablet for 8 weeks. Participant is then co-administered MK-0524A 2 g + simvastatin 40 mg for 8 weeks.
  Interventions: Drug: Comparator: simvastatin; Drug: MK-0524A; Drug: Placebo; Drug: MK-0524B
- Sequence 4: MK-0524A 2g+Simvastatin 40mg →MK-0524B 1.8g/40mg (Experimental): After a 2-week placebo run-in, participants will be co-administered MK-0524A 1g + simvastatin 40 mg for 4 weeks, then co-administration MK-0524A 2g +simvastatin 40 mg for 8 weeks. Participant then receives MK-0524B 1.8 g/40 mg combination tablet for 8 weeks.
  Interventions: Drug: Comparator: simvastatin; Drug: MK-0524A; Drug: Placebo; Drug: MK-0524B

INTERVENTIONS:
Drug: Comparator: simvastatin
  Other Names: Zocor®; MK0733
Drug: MK-0524A — Extended-release(ER) niacin/Laropiprant (MK-0524) Combination tablet
Drug: Placebo
Drug: MK-0524B

SUMMARY:
This is a 20-week clinical trial in participants with primary hypercholesterolemia or mixed dyslipidemia to demonstrate the effect of MK-0524B compared to MK-0524A + Simvastatin on lipid values.

ELIGIBILITY:
Inclusion Criteria:

* has primary hypercholesterolemia or mixed dyslipidemia based on medical history (previous diagnosis), historic lipid values, or as otherwise determined through optional lipid measurements at screening visit
* meets one of the following triglyceride (TG) criteria:

  1. is on niacin, statin, or fibrate and has TG <500 mg/dL at or within 6 months of washout
  2. is not on any lipid altering therapy or is on lipid altering therapy other than niacin, statin, or fibrate and has TG <600 mg/dL at or within 6 months of screening

Exclusion Criteria:

* is high risk (coronary heart disease [CHD] or CHD risk equivalent) AND is on a statin
* is pregnant or breast-feeding, or expecting to conceive during the study including the 14-day post study follow-up
* has Type 1 or Type 2 diabetes mellitus and is on statin therapy, is poorly controlled, is newly diagnosed (within 3 months of Visit 1), has recently experienced repeated hypoglycemia or unstable glycemic control or is taking new or recently adjusted anti-diabetic medications (with the exception of +/- 10 units of insulin) within 3 months of Visit 1
* has the following conditions: chronic heart failure, uncontrolled/unstable cardiac arrhythmias, unstable hypertension, active or chronic hepatobiliary disorder or hepatic disease, human immunodeficiency virus (HIV) positive, gout (within 1 year)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2414 (Actual)
Dates: Start 2007-06-15 (Actual); Primary Completion 2008-06-16 (Actual); Study Completion 2008-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis Link — http://www.merck.com/clinical-trials/study.html?id=0524B-063&kw=0524B-063&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants completed a 6-8 week washout then completed a 2-week placebo run-in prior to the start of active treatment. Includes 6 participants who had an adverse event that began during the placebo run-in but did not lead to discontinuation until after randomization in Period I or II.
Period: Precrossover: Periods I/II (Weeks 1-12)
Arm/Group | Sequence 1: MK-0524B 1.8g/20mg→MK-0524A 2g+Simvastatin 20mg | Sequence 2: MK-0524A 2g+Simvastatin 20mg →MK-0524B 1.8g/20mg | Sequence 3: MK-0524B 1.8g/40mg→MK-0524A 2g+Simvastatin 40mg | Sequence 4: MK-0524A 2g+Simvastatin 40mg →MK-0524B 1.8g/40mg
Started | 610 | 602 | 597 | 605
Completed | 472 | 440 | 440 | 465
Not Completed | 138 | 162 | 157 | 140
Not completed — Clinical Adverse Event | 96 | 99 | 98 | 87
Not completed — Laboratory Adverse Event | 0 | 4 | 4 | 4
Not completed — Lost to Follow-up | 12 | 9 | 9 | 11
Not completed — Other | 4 | 6 | 9 | 5
Not completed — Participant moved | 0 | 4 | 2 | 1
Not completed — Withdrawal by Subject | 24 | 33 | 30 | 25
Not completed — Protocol Violation | 2 | 7 | 5 | 7
Period: Crossover: Period III (Weeks 13-20)
Arm/Group | Sequence 1: MK-0524B 1.8g/20mg→MK-0524A 2g+Simvastatin 20mg | Sequence 2: MK-0524A 2g+Simvastatin 20mg →MK-0524B 1.8g/20mg | Sequence 3: MK-0524B 1.8g/40mg→MK-0524A 2g+Simvastatin 40mg | Sequence 4: MK-0524A 2g+Simvastatin 40mg →MK-0524B 1.8g/40mg
Started | 472 | 440 | 440 | 465
Completed | 447 | 419 | 420 | 447
Not Completed | 25 | 21 | 20 | 18
Not completed — Clinical Adverse Event | 12 | 13 | 12 | 10
Not completed — Laboratory Adverse Event | 3 | 1 | 2 | 2
Not completed — Lost to Follow-up | 1 | 2 | 1 | 1
Not completed — Other | 5 | 0 | 2 | 2
Not completed — Participant moved | 1 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 1 | 3
Not completed — Protocol Violation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1: MK-0524B 1.8g/20mg→MK-0524A 2g+Simvastatin 20mg | Sequence 2: MK-0524A 2g+Simvastatin 20mg →MK-0524B 1.8g/20mg | Sequence 3: MK-0524B 1.8g/40mg→MK-0524A 2g+Simvastatin 40mg | Sequence 4: MK-0524A 2g+Simvastatin 40mg →MK-0524B 1.8g/40mg | Total
Number analyzed (Participants) | 610 | 602 | 597 | 605 | 2414
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 491 | 470 | 468 | 477 | 1906
  >=65 years | 119 | 132 | 129 | 128 | 508
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 325 | 334 | 313 | 316 | 1288
  Male | 285 | 268 | 284 | 289 | 1126

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C)
Description: Blood samples taken at baseline (Week 4 for Period II; Week 12 for Period III) and after 8 weeks of treatment during each period to determine the LDL-C levels. The change from baseline after 8 weeks of treatment was recorded.
Time Frame: Baseline (Week 4 for Period II; Week 12 for Period III) and after 8 weeks of treatment during each period (Week 12 for Period II and Week 20 for Period III)
Population: Participants who completed the study and had respective endpoint data available at baseline and end of each treatment period. End of period value was defined as measurements collected on the same date as the corresponding end of period visit date. Results were reported by dose of study drug taken and not by randomly assigned sequence.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Groups:
- MK-0524B 1.8g/20mg: Participants who received MK-0524B 1.8g/20mg for 8 weeks in either Period II or Period III regardless of randomly assigned sequence.
- MK-0524A 2g+Simvastatin 20mg: Participants who received MK-0524A 2g+Simvastatin 20mg for 8 weeks in either Period II or Period III regardless of randomly assigned sequence.
- MK-0524B 1.8g/40mg: Participants who received MK-0524B 1.8g/40mg for 8 weeks in either Period II or Period III treatment period regardless of randomly assigned sequence.
- MK-0524A 2g+Simvastatin 40mg: Participants who received MK-0524A 2g+Simvastatin 40mg for 8 weeks in either Period II or Period III regardless of randomly assigned sequence.
Arm/Group | MK-0524B 1.8g/20mg | MK-0524A 2g+Simvastatin 20mg | MK-0524B 1.8g/40mg | MK-0524A 2g+Simvastatin 40mg
Number analyzed (Participants) | 844 | 844 | 843 | 843
Percentage Change | -44.6 [-45.3 to -43.8] | -46.9 [-47.7 to -46.2] | -48.9 [-49.7 to -48.2] | -50.4 [-51.1 to -49.7]
Statistical Analysis 1: Comparison: MK-0524B 1.8g/20mg vs MK-0524A 2g+Simvastatin 20mg; Test type: Non-Inferiority or Equivalence — Clinical equivalence LDL-C reduction was established if the 95% CI for the difference between these two treatments in percent change from baseline in LDL-C fell within ±3%; ANOVA; Factors for sequence, participant within sequence, period and treatment; Difference in Least squares mean = 2.4, 95% CI 2-sided [1.3 to 3.4]
Statistical Analysis 2: Comparison: MK-0524B 1.8g/40mg vs MK-0524A 2g+Simvastatin 40mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Factors for sequence, participant within sequence, period and treatment; Difference in Least Squares Mean = 1.4, 95% CI 2-sided [0.4 to 2.4]

2. Secondary Outcome: Percentage Change From Baseline in High-density Lipoprotein Cholesterol (HDL-C)
Description: Blood samples taken at baseline (Week 4 for Period II; Week 12 for Period III) and after 8 weeks of treatment during each period to determine the HDL-C levels. The change from baseline after 8 weeks of treatment was recorded.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | MK-0524B 1.8g/20mg | MK-0524A 2g+Simvastatin 20mg | MK-0524B 1.8g/40mg | MK-0524A 2g+Simvastatin 40mg
Number analyzed (Participants) | 845 | 845 | 845 | 845
Percentage Change | 27.4 [26.5 to 28.2] | 27.6 [26.7 to 28.4] | 27.7 [26.9 to 28.4] | 28.5 [27.8 to 29.2]
Statistical Analysis 1: Comparison: MK-0524B 1.8g/20mg vs MK-0524A 2g+Simvastatin 20mg; Test type: Non-Inferiority or Equivalence — Clinical equivalence HDL-C reduction was established if the 95% CI for the difference between these two treatments in percent change from baseline in LDL-C fell within ±4%; ANOVA; Factors for sequence, participant within sequence, period and treatment; Difference in Least Squares Mean = -0.2, 95% CI 2-sided [-1.4 to 1.0]
Statistical Analysis 2: Comparison: MK-0524B 1.8g/40mg vs MK-0524A 2g+Simvastatin 40mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; Factors for sequence, participant within sequence, period and treatment; Difference in Least Squares Mean = -0.8, 95% CI 2-sided [-1.9 to 0.2]

3. Secondary Outcome: Percentage of Participants With Consecutive Elevations in Alanine Aminotransferase (ALT) and/or Aspartate Aminotransferase (AST) of >=3 x Upper Limit of Normal (ULN)
Description: Participants had AST and ALT levels assessed during Period I (4 weeks ) throughout each 8 week treatment period (20 weeks total). Participants who had an assessment of either AST or ALT that was 3 x ULN or greater were recorded. The AST ULNs for males and females were 43 U/L and 36 U/L, respectively. The ALT ULNs for males and females were 40 U/L and 33 U/L, respectively.
Time Frame: up 20 weeks (12 weeks in Period I/II and 8 weeks in Period III)
Population: All participants who received at least 1 dose of study drug. Safety analysis was based on the experiences accumulated during Periods I/II combined (pre-crossover), where the study follows a parallel design. A separate safety analysis was performed for Period III (post-crossover).
Measure: Number; unit: Percentage of Participants
Groups:
- Sequence 1: MK-0524B 1.8g/20mg: Participants who received MK-0524B 0.9g/20mg and MK-0524B 1.8g/20mg during Periods I/II
- Sequence 2: MK-0524A 2g+Simvastatin 20mg: Participants who received MK-0524A 1g + Simvastatin 20mg and MK-0524A 2g+ Simvastatin 20mg during Periods I/II.
- Sequence 1: MK-0524A 2g+Simvastatin 20mg: Participants who received MK-0524A 1g + Simvastatin 20mg and MK-0524A 2g+ Simvastatin 20mg during Period III
- Sequence 2: MK-0524B 1.8g/20mg: Participants who received MK-0524B 1.8g/20mg during Periods III
- Sequence 3: MK-0524B 1.8g/40mg: Participants who received MK-0524B 0.9g/40mg and MK-0524B 1.8g/40mg during Periods I/II
- Sequence 4: MK-0524A 2g+Simvastatin 40mg: Participants who received MK-0524A 1g + Simvastatin 40mg and MK-0524A 2g+ Simvastatin 40mg during Periods I/II.
- Sequence 3: MK-0524A 2g+Simvastatin 40mg: Participants who received MK-0524A 1g + Simvastatin 40mg and MK-0524A 2g+ Simvastatin 40mg during Period III
- Sequence 4: MK-0524B 1.8g/40mg: Participants who received MK-0524B 1.8g/40mg during Periods III
Arm/Group | Sequence 1: MK-0524B 1.8g/20mg | Sequence 2: MK-0524A 2g+Simvastatin 20mg | Sequence 1: MK-0524A 2g+Simvastatin 20mg | Sequence 2: MK-0524B 1.8g/20mg | Sequence 3: MK-0524B 1.8g/40mg | Sequence 4: MK-0524A 2g+Simvastatin 40mg | Sequence 3: MK-0524A 2g+Simvastatin 40mg | Sequence 4: MK-0524B 1.8g/40mg
Number analyzed (Participants) | 588 | 580 | 469 | 437 | 568 | 592 | 438 | 464
Percentage of Participants | 0.3 | 0.5 | 0.6 | 0.9 | 0.7 | 1.0 | 0.5 | 0.2
Statistical Analysis 1: Comparison: Sequence 1: MK-0524B 1.8g/20mg vs Sequence 2: MK-0524A 2g+Simvastatin 20mg; Periods I/II; Test type: Superiority or Other; p = 0.685, Fisher Exact; Difference in Percentage = -0.2, 95% CI 2-sided [-1.2 to 0.8] — Wilson's Method
Statistical Analysis 2: Comparison: Sequence 1: MK-0524A 2g+Simvastatin 20mg vs Sequence 2: MK-0524B 1.8g/20mg; Period III; Test type: Superiority or Other; Difference in Percentage = -0.3, 95% CI 2-sided [-1.8 to 1.1] — Wilson's Method
Statistical Analysis 3: Comparison: Sequence 3: MK-0524B 1.8g/40mg vs Sequence 4: MK-0524A 2g+Simvastatin 40mg; Periods I/II; Test type: Superiority or Other; p = 0.753, Fisher Exact; Difference in Percentage = -0.3, 95% CI 2-sided [-1.6 to 0.9] — Wilson's Method
Statistical Analysis 4: Comparison: Sequence 3: MK-0524A 2g+Simvastatin 40mg vs Sequence 4: MK-0524B 1.8g/40mg; Period III; Test type: Superiority or Other; Difference in Percentage = 0.2, 95% CI 2-sided [-0.8 to 1.4] — Wilson's Method

4. Secondary Outcome: Percentage of Participants With Creatine Kinase (CK) >=10 x ULN
Description: Participants had CK levels assessed during Period I (4 weeks ) throughout each 8 week treatment period (20 weeks total). Participants who had an assessment of CK that was 10 x ULN or greater were recorded. The ULNs for males and females were 207 U/L and 169 U/L, respectively.
Time Frame: up 20 weeks (12 weeks in Period I/II and 8 weeks in Period III)
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 1.8g/20mg | Sequence 2: MK-0524A 2g+Simvastatin 20mg | Sequence 1: MK-0524A 2g+Simvastatin 20mg | Sequence 2: MK-0524B 1.8g/20mg | Sequence 3: MK-0524B 1.8g/40mg | Sequence 4: MK-0524A 2g+Simvastatin 40mg | Sequence 3: MK-0524A 2g+Simvastatin 40mg | Sequence 4: MK-0524B 1.8g/40mg
Number analyzed (Participants) | 588 | 580 | 469 | 437 | 568 | 592 | 438 | 464
Percentage of Participants | 0.0 | 0.0 | 0.4 | 0.0 | 0.4 | 0.2 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Sequence 1: MK-0524B 1.8g/20mg vs Sequence 2: MK-0524A 2g+Simvastatin 20mg; Periods I/II; Test type: Superiority or Other; Fisher Exact; Difference in Percentage = 0.0, 95% CI 2-sided [-0.7 to 0.6] — Wilson's Method
Statistical Analysis 2: Comparison: Sequence 1: MK-0524A 2g+Simvastatin 20mg vs Sequence 2: MK-0524B 1.8g/20mg; Period III; Test type: Superiority or Other; Difference in Percentage = 0.4, 95% CI 2-sided [-0.5 to 1.5] — Wilson's Method
Statistical Analysis 3: Comparison: Sequence 3: MK-0524B 1.8g/40mg vs Sequence 4: MK-0524A 2g+Simvastatin 40mg; Periods I/II; Test type: Superiority or Other; p = 0.617, Fisher Exact; Difference in Percentage = 0.2, 95% CI 2-sided [-0.6 to 1.1] — Wilson's Method
Statistical Analysis 4: Comparison: Sequence 3: MK-0524A 2g+Simvastatin 40mg vs Sequence 4: MK-0524B 1.8g/40mg; Period III; Test type: Superiority or Other; Difference in Percentage = 0.0, 95% CI 2-sided [-0.8 to 0.9] — Wilson's Method

5. Secondary Outcome: Percentage of Participants With CK >=10 x ULN With Muscle Symptoms
Description: Participants had CK levels assessed during Period I (4 weeks ) throughout each 8 week treatment period (20 weeks total). Participants who had an assessment of CK that was 10 x ULN or greater and had associated muscle symptoms present within +/- 7 days were recorded. The ULNs for males and females were 207 U/L and 169 U/L, respectively.
Time Frame: up 20 weeks (12 weeks in Period I/II and 8 weeks in Period III)
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 1.8g/20mg | Sequence 2: MK-0524A 2g+Simvastatin 20mg | Sequence 1: MK-0524A 2g+Simvastatin 20mg | Sequence 2: MK-0524B 1.8g/20mg | Sequence 3: MK-0524B 1.8g/40mg | Sequence 4: MK-0524A 2g+Simvastatin 40mg | Sequence 3: MK-0524A 2g+Simvastatin 40mg | Sequence 4: MK-0524B 1.8g/40mg
Number analyzed (Participants) | 588 | 580 | 469 | 437 | 568 | 592 | 438 | 464
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Sequence 1: MK-0524B 1.8g/20mg vs Sequence 2: MK-0524A 2g+Simvastatin 20mg; Periods I/II; Test type: Superiority or Other; Fisher Exact; Difference in Percentage = 0.0, 95% CI 2-sided [-0.7 to 0.6] — Wilson's Method
Statistical Analysis 2: Comparison: Sequence 1: MK-0524A 2g+Simvastatin 20mg vs Sequence 2: MK-0524B 1.8g/20mg; Period III; Test type: Superiority or Other; Difference in Percentage = 0.0, 95% CI 2-sided [-0.9 to 0.8] — Wilson's Method
Statistical Analysis 3: Comparison: Sequence 3: MK-0524B 1.8g/40mg vs Sequence 4: MK-0524A 2g+Simvastatin 40mg; Periods I/II; Test type: Superiority or Other; Fisher Exact; Difference in Percentage = 0.0, 95% CI 2-sided [-0.6 to 0.7] — Wilson's Method
Statistical Analysis 4: Comparison: Sequence 3: MK-0524A 2g+Simvastatin 40mg vs Sequence 4: MK-0524B 1.8g/40mg; Period III; Test type: Superiority or Other; Difference in Percentage = 0.0, 95% CI 2-sided [-0.8 to 0.9] — Wilson's Method

6. Secondary Outcome: Percentage of Participants With CK >=10 x ULN With Muscle Symptoms - Drug Related
Description: Participants had CK levels assessed during Period I (4 weeks ) throughout each 8 week treatment period (20 weeks total). Participants who had an assessment of CK that was 10 x ULN or greater and had associated muscle symptoms present within +/- 7 days that were reported as at least possibly related to study drug were recorded. The ULNs for males and females were 207 U/L and 169 U/L, respectively.
Time Frame: up 20 weeks (12 weeks in Period I/II and 8 weeks in Period III)
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 1.8g/20mg | Sequence 2: MK-0524A 2g+Simvastatin 20mg | Sequence 1: MK-0524A 2g+Simvastatin 20mg | Sequence 2: MK-0524B 1.8g/20mg | Sequence 3: MK-0524B 1.8g/40mg | Sequence 4: MK-0524A 2g+Simvastatin 40mg | Sequence 3: MK-0524A 2g+Simvastatin 40mg | Sequence 4: MK-0524B 1.8g/40mg
Number analyzed (Participants) | 588 | 580 | 469 | 437 | 568 | 592 | 438 | 464
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Sequence 1: MK-0524B 1.8g/20mg vs Sequence 2: MK-0524A 2g+Simvastatin 20mg; Periods I/II; Test type: Superiority or Other; Fisher Exact; Difference in Percentage = 0.0, 95% CI 2-sided [-0.7 to 0.6] — Wilson's Method
Statistical Analysis 2: Comparison: Sequence 1: MK-0524A 2g+Simvastatin 20mg vs Sequence 2: MK-0524B 1.8g/20mg; Period III; Test type: Superiority or Other; Difference in Percentage = 0.0, 95% CI 2-sided [-0.9 to 0.8] — Wilson's Method
Statistical Analysis 3: Comparison: Sequence 3: MK-0524B 1.8g/40mg vs Sequence 4: MK-0524A 2g+Simvastatin 40mg; Periods I/II; Test type: Superiority or Other; Fisher Exact; Difference in Percentage = 0.0, 95% CI 2-sided [-0.6 to 0.7] — Wilson's Method
Statistical Analysis 4: Comparison: Sequence 3: MK-0524A 2g+Simvastatin 40mg vs Sequence 4: MK-0524B 1.8g/40mg; Period III; Test type: Superiority or Other; Difference in Percentage = 0.0, 95% CI 2-sided [-0.8 to 0.9] — Wilson's Method

7. Secondary Outcome: Percentage of Participants With New Diagnosis of Impaired Fasting Blood Glucose
Description: Participants had fasting glucose levels assessed during Period I (4 weeks ) throughout each 8 week treatment period (20 weeks total). Participants who had the new diagnosis of impaired fasting blood glucose were recorded. A pre-defined set of MedDRA terms was used to identify participants whose glycemic status became 'impaired' during the course of treatment (from clinical adverse experience reports). The MedDRA terms were as follows: blood glucose increased, blood glucose abnormal, glucose tolerance decreased, glucose tolerance test abnormal, carbohydrate tolerance decreased, glucose tolerance impaired, hyperglycaemia, impaired fasting glucose, impaired insulin secretion, metabolic syndrome, insulin resistance, insulin resistance syndrome.
Time Frame: up 20 weeks (12 weeks in Period I/II and 8 weeks in Period III)
Population: All participants who had normal fasting blood glucose levels at baseline and who received at least 1 dose of study drug. Safety analysis was based on the experiences accumulated during Periods I/II combined (pre-crossover), where the study follows a parallel design. A separate safety analysis was performed for Period III (post-crossover).
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 1.8g/20mg | Sequence 2: MK-0524A 2g+Simvastatin 20mg | Sequence 1: MK-0524A 2g+Simvastatin 20mg | Sequence 2: MK-0524B 1.8g/20mg | Sequence 3: MK-0524B 1.8g/40mg | Sequence 4: MK-0524A 2g+Simvastatin 40mg | Sequence 3: MK-0524A 2g+Simvastatin 40mg | Sequence 4: MK-0524B 1.8g/40mg
Number analyzed (Participants) | 484 | 473 | 468 | 483 | 365 | 343 | 345 | 372
Percentage of Participants | 0.0 | 0.2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Sequence 1: MK-0524B 1.8g/20mg vs Sequence 2: MK-0524A 2g+Simvastatin 20mg; Periods I/II; Test type: Superiority or Other; p = 0.497, Fisher Exact; Difference in Percentage = -0.2, 95% CI 2-sided [-0.9 to 0.5]

8. Secondary Outcome: Percentage of Participants With New Diagnosis of Diabetes
Description: Participants who with newly diagnosed of diabetes were recorded. A participant was classified as having new onset diabetes if they experienced an adverse Event (AE) related to a diagnosis of diabetes (based on a pre-defined set of Medical Dictionary for Regulatory Activities [MedDRA] terms), or if they started taking an anti-diabetic medication during the course of the study. The MedDRA terms were as follows: diabetes mellitus, diabetes mellitus insulin-dependent, diabetes mellitus non-insulin dependent, insulin-requiring type II diabetes mellitus, insulin resistant diabetes, diabetes with hyperosmolarity, latent autoimmune diabetes in adults.
Time Frame: up 20 weeks (12 weeks in Period I/II and 8 weeks in Period III)
Population: All participants without diabetes at baseline and who received at least 1 dose of study drug. Safety analysis was based on the experiences accumulated during Periods I/II combined (pre-crossover), where the study follows a parallel design. A separate safety analysis was performed for Period III (post-crossover).
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 1.8g/20mg | Sequence 2: MK-0524A 2g+Simvastatin 20mg | Sequence 1: MK-0524A 2g+Simvastatin 20mg | Sequence 2: MK-0524B 1.8g/20mg | Sequence 3: MK-0524B 1.8g/40mg | Sequence 4: MK-0524A 2g+Simvastatin 40mg | Sequence 3: MK-0524A 2g+Simvastatin 40mg | Sequence 4: MK-0524B 1.8g/40mg
Number analyzed (Participants) | 554 | 551 | 427 | 404 | 545 | 545 | 404 | 422
Percentage of Participants | 0.4 | 0.7 | 0.5 | 0.7 | 0.6 | 0.4 | 0.7 | 0.5
Statistical Analysis 1: Comparison: Sequence 1: MK-0524B 1.8g/20mg vs Sequence 2: MK-0524A 2g+Simvastatin 20mg; Periods I/II; Test type: Superiority or Other; p = 0.449, Fisher Exact; Difference in Percentage = -0.3, 95% CI 2-sided [-1.4 to 0.6] — Wilson's Method
Statistical Analysis 2: Comparison: Sequence 1: MK-0524A 2g+Simvastatin 20mg vs Sequence 2: MK-0524B 1.8g/20mg; Period III; Test type: Superiority or Other; Difference in Percentage = -0.3, 95% CI 2-sided [-1.6 to 0.9] — Wilson's Method
Statistical Analysis 3: Comparison: Sequence 3: MK-0524B 1.8g/40mg vs Sequence 4: MK-0524A 2g+Simvastatin 40mg; Period I/II; Test type: Superiority or Other; p = 0.685, Fisher Exact; Difference in Percentage = 0.2, 95% CI 2-sided [-0.8 to 1.2] — Wilson's Method
Statistical Analysis 4: Comparison: Sequence 3: MK-0524A 2g+Simvastatin 40mg vs Sequence 4: MK-0524B 1.8g/40mg; Period III; Test type: Superiority or Other; Difference in Percentage = 0.3, 95% CI 2-sided [-1.0 to 1.6] — Wilson's Method

9. Secondary Outcome: Percentage of Participants With Worsening of the Pre-existing Conditions of Diabetes in Participants With Diabetes at Baseline
Description: Participants with diabetes at baseline and who experienced a worsening of the diabetes identified through adverse event reports using a pre-defined set of terms and/or increasing dose/adding a new anti-diabetic medication.
Time Frame: up 20 weeks (12 weeks in Period I/II and 8 weeks in Period III)
Population: All participants with diabetes at baseline and who received at least 1 dose of study drug. Safety analysis was based on the experiences accumulated during Periods I/II combined (pre-crossover), where the study follows a parallel design. A separate safety analysis was performed for Period III (post-crossover).
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 1.8g/20mg | Sequence 2: MK-0524A 2g+Simvastatin 20mg | Sequence 1: MK-0524A 2g+Simvastatin 20mg | Sequence 2: MK-0524B 1.8g/20mg | Sequence 3: MK-0524B 1.8g/40mg | Sequence 4: MK-0524A 2g+Simvastatin 40mg | Sequence 3: MK-0524A 2g+Simvastatin 40mg | Sequence 4: MK-0524B 1.8g/40mg
Number analyzed (Participants) | 56 | 51 | 45 | 36 | 52 | 60 | 36 | 43
Percentage of Participants | 1.8 | 15.7 | 4.4 | 8.3 | 3.8 | 8.3 | 8.3 | 11.6
Statistical Analysis 1: Comparison: Sequence 1: MK-0524B 1.8g/20mg vs Sequence 2: MK-0524A 2g+Simvastatin 20mg; Periods I/II; Test type: Superiority or Other; p = 0.020, Fisher Exact; Difference in Percentage = -1.2, 95% CI 2-sided [-2.4 to -0.2] — Wilson's Method
Statistical Analysis 2: Comparison: Sequence 1: MK-0524A 2g+Simvastatin 20mg vs Sequence 2: MK-0524B 1.8g/20mg; Period III; Test type: Superiority or Other; Difference in Percentage = -0.3, 95% CI 2-sided [-1.6 to 0.9] — Wilson's Method
Statistical Analysis 3: Comparison: Sequence 3: MK-0524B 1.8g/40mg vs Sequence 4: MK-0524A 2g+Simvastatin 40mg; Periods I/II; Test type: Superiority or Other; p = 0.452, Fisher Exact; Difference in Percentage = -0.5, 95% CI 2-sided [-1.6 to 0.5] — Wilson's Method
Statistical Analysis 4: Comparison: Sequence 3: MK-0524A 2g+Simvastatin 40mg vs Sequence 4: MK-0524B 1.8g/40mg; Period III; Test type: Superiority or Other; Difference in Percentage = -0.4, 95% CI 2-sided [-1.9 to 1.0] — Wilson's Method

10. Secondary Outcome: Percentage of Participants With a Confirmed Adjudicated Cardiovascular Event
Description: Select serious adverse cardiovascular events and all-cause mortality that occurred during the treatment phase of the study were adjudicated by an expert committee external to the sponsor. Those events confirmed by the committee as cardiovascular events were recorded
Time Frame: up 20 weeks (12 weeks in Period I/II and 8 weeks in Period III)
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 1.8g/20mg | Sequence 2: MK-0524A 2g+Simvastatin 20mg | Sequence 1: MK-0524A 2g+Simvastatin 20mg | Sequence 2: MK-0524B 1.8g/20mg | Sequence 3: MK-0524B 1.8g/40mg | Sequence 4: MK-0524A 2g+Simvastatin 40mg | Sequence 3: MK-0524A 2g+Simvastatin 40mg | Sequence 4: MK-0524B 1.8g/40mg
Number analyzed (Participants) | 610 | 602 | 472 | 440 | 597 | 605 | 440 | 465
Percentage of Participants | 0.0 | 0.0 | 0.2 | 0.0 | 0.2 | 0.0 | 0.2 | 0.0
Statistical Analysis 1: Comparison: Sequence 1: MK-0524B 1.8g/20mg vs Sequence 2: MK-0524A 2g+Simvastatin 20mg; Periods I/II; Test type: Superiority or Other; Difference in Percentage = 0.0, 95% CI 2-sided [-0.6 to 0.6] — Wilson's Method
Statistical Analysis 2: Comparison: Sequence 1: MK-0524A 2g+Simvastatin 20mg vs Sequence 2: MK-0524B 1.8g/20mg; Period III; Test type: Superiority or Other; Difference in Percentage = 0.2, 95% CI 2-sided [-0.7 to 1.2] — Wilson's Method
Statistical Analysis 3: Comparison: Sequence 3: MK-0524B 1.8g/40mg vs Sequence 4: MK-0524A 2g+Simvastatin 40mg; Periods I/II; Test type: Superiority or Other; Difference in Percentage = 0.2, 95% CI 2-sided [-0.5 to 0.9] — Wilson's Method
Statistical Analysis 4: Comparison: Sequence 3: MK-0524A 2g+Simvastatin 40mg vs Sequence 4: MK-0524B 1.8g/40mg; Period III; Test type: Superiority or Other; Difference in Percentage = 0.2, 95% CI 2-sided [-0.6 to 1.3] — Wilson's Method

11. Secondary Outcome: Percentage of Participants Who Experience at Least 1 Clinical Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. A clinical AE was an AE reported as a result of a clinical examination or reported by the participant.
Time Frame: up 20 weeks (12 weeks in Period I/II and 8 weeks in Period III)
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 1.8g/20mg | Sequence 2: MK-0524A 2g+Simvastatin 20mg | Sequence 1: MK-0524A 2g+Simvastatin 20mg | Sequence 2: MK-0524B 1.8g/20mg | Sequence 3: MK-0524B 1.8g/40mg | Sequence 4: MK-0524A 2g+Simvastatin 40mg | Sequence 3: MK-0524A 2g+Simvastatin 40mg | Sequence 4: MK-0524B 1.8g/40mg
Number analyzed (Participants) | 610 | 602 | 472 | 440 | 597 | 605 | 440 | 465
Percentage of Participants | 67.5 | 68.9 | 35.6 | 37.5 | 67.5 | 67.4 | 32.3 | 35.1
Statistical Analysis 1: Comparison: Sequence 1: MK-0524B 1.8g/20mg vs Sequence 2: MK-0524A 2g+Simvastatin 20mg; Periods I/II; Test type: Superiority or Other; Difference in Percentage = -1.4, 95% CI 2-sided [-6.6 to 3.8] — Wilson's Score Method
Statistical Analysis 2: Comparison: Sequence 1: MK-0524A 2g+Simvastatin 20mg vs Sequence 2: MK-0524B 1.8g/20mg; Period III; Test type: Superiority or Other; Difference in Percentage = -1.9, 95% CI 2-sided [-8.1 to 4.3] — Wilson's Score Method
Statistical Analysis 3: Comparison: Sequence 3: MK-0524B 1.8g/40mg vs Sequence 4: MK-0524A 2g+Simvastatin 40mg; Periods I/II; Test type: Superiority or Other; Difference in Percentage = 0.1, 95% CI 2-sided [-5.2 to 5.3] — Wilson's Score Method
Statistical Analysis 4: Comparison: Sequence 3: MK-0524A 2g+Simvastatin 40mg vs Sequence 4: MK-0524B 1.8g/40mg; Period III; Test type: Superiority or Other; Difference in Percentage = -2.8, 95% CI 2-sided [-8.9 to 3.4] — Wilson's Score Method

12. Secondary Outcome: Percentage of Participants Who Experience at Least 1 Laboratory AE
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. A laboratory AE was an AE reported as a result of a laboratory assessment or test
Time Frame: up 20 weeks (12 weeks in Period I/II and 8 weeks in Period III)
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 1.8g/20mg | Sequence 2: MK-0524A 2g+Simvastatin 20mg | Sequence 1: MK-0524A 2g+Simvastatin 20mg | Sequence 2: MK-0524B 1.8g/20mg | Sequence 3: MK-0524B 1.8g/40mg | Sequence 4: MK-0524A 2g+Simvastatin 40mg | Sequence 3: MK-0524A 2g+Simvastatin 40mg | Sequence 4: MK-0524B 1.8g/40mg
Number analyzed (Participants) | 610 | 602 | 472 | 440 | 597 | 605 | 440 | 465
Percentage of Participants | 3.9 | 4.2 | 5.9 | 3.6 | 6.2 | 4.6 | 5.9 | 3.9
Statistical Analysis 1: Comparison: Sequence 1: MK-0524B 1.8g/20mg vs Sequence 2: MK-0524A 2g+Simvastatin 20mg; Periods I/II; Test type: Superiority or Other; Difference in Percentage = -0.2, 95% CI 2-sided [-2.5 to 2.1] — Wilson's Score Method
Statistical Analysis 2: Comparison: Sequence 1: MK-0524A 2g+Simvastatin 20mg vs Sequence 2: MK-0524B 1.8g/20mg; Period III; Test type: Superiority or Other; Difference in Percentage = 2.3, 95% CI 2-sided [-0.5 to 5.2] — Wilson's Score Method
Statistical Analysis 3: Comparison: Sequence 3: MK-0524B 1.8g/40mg vs Sequence 4: MK-0524A 2g+Simvastatin 40mg; Periods I/II; Test type: Superiority or Other; Difference in Percentage = 1.6, 95% CI 2-sided [-1.0 to 4.2] — Wilson's Score Method
Statistical Analysis 4: Comparison: Sequence 3: MK-0524A 2g+Simvastatin 40mg vs Sequence 4: MK-0524B 1.8g/40mg; Period III; Test type: Superiority or Other; Difference in Percentage = 2.0, 95% CI 2-sided [-0.8 to 5.0] — Wilson's Score Method

13. Secondary Outcome: Percentage of Participants Who Were Discontinued From the Study Due to a Clinical AE
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. A clinical AE was an AE reported as a result of a clinical examination or reported by the participant. Participants who were discontinued from the study due to a clinical AE were recorded.
Time Frame: up 20 weeks (12 weeks in Period I/II and 8 weeks in Period III)
Population: All participants who received at least 1 dose of study drug. Safety analysis was based on the experiences accumulated during Periods I/II combined, where the study follows a parallel design. A separate safety analysis was performed for Period III (post-crossover). Excludes 6 participants who had an AE that began during the placebo run-in.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 1.8g/20mg | Sequence 2: MK-0524A 2g+Simvastatin 20mg | Sequence 1: MK-0524A 2g+Simvastatin 20mg | Sequence 2: MK-0524B 1.8g/20mg | Sequence 3: MK-0524B 1.8g/40mg | Sequence 4: MK-0524A 2g+Simvastatin 40mg | Sequence 3: MK-0524A 2g+Simvastatin 40mg | Sequence 4: MK-0524B 1.8g/40mg
Number analyzed (Participants) | 610 | 602 | 472 | 440 | 597 | 605 | 440 | 465
Percentage of Participants | 15.9 | 15.9 | 1.9 | 2.7 | 16.4 | 14.4 | 2.5 | 1.5

14. Secondary Outcome: Percentage of Participants Who Were Discontinued From the Study Due to a Laboratory AE
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. A laboratory AE was an AE reported as a result of a laboratory assessment or test. Participants who were discontinued from the study due to a laboratory AE were recorded.
Time Frame: up 20 weeks (12 weeks in Period I/II and 8 weeks in Period III)
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 1.8g/20mg | Sequence 2: MK-0524A 2g+Simvastatin 20mg | Sequence 1: MK-0524A 2g+Simvastatin 20mg | Sequence 2: MK-0524B 1.8g/20mg | Sequence 3: MK-0524B 1.8g/40mg | Sequence 4: MK-0524A 2g+Simvastatin 40mg | Sequence 3: MK-0524A 2g+Simvastatin 40mg | Sequence 4: MK-0524B 1.8g/40mg
Number analyzed (Participants) | 610 | 602 | 472 | 440 | 597 | 605 | 440 | 465
Percentage of Participants | 0.0 | 0.7 | 0.6 | 0.2 | 0.7 | 0.8 | 0.5 | 0.2

15. Secondary Outcome: Percentage of Participants Who Experience at Least 1 Hepatitis-related Non-serious Clinical AE
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. Non-serious Hepatitis-related AEs were identified by a collective review using the following pre-specified set of preferred terms: cholestasis, hepatic necrosis, hepatocellular damage, cytolytic hepatitis, hepatitis, hepatomegaly, jaundice, hepatic failure, hepatitis cholestatic, jaundice cholestatic, hepatitis fulminant, hyperbilirubinaemia, jaundice hepatocellular, ocular icterus, yellow skin, hepatic function abnormal, acute hepatic failure, subacute hepatic failure, hepatitis acute, hepatitis toxic, hepatotoxicity, and mixed hepatocellular-cholestatic injury.
Time Frame: up 20 weeks (12 weeks in Period I/II and 8 weeks in Period III)
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Sequence 1: MK-0524B 1.8g/20mg | Sequence 2: MK-0524A 2g+Simvastatin 20mg | Sequence 1: MK-0524A 2g+Simvastatin 20mg | Sequence 2: MK-0524B 1.8g/20mg | Sequence 3: MK-0524B 1.8g/40mg | Sequence 4: MK-0524A 2g+Simvastatin 40mg | Sequence 3: MK-0524A 2g+Simvastatin 40mg | Sequence 4: MK-0524B 1.8g/40mg
Number analyzed (Participants) | 610 | 602 | 472 | 440 | 597 | 605 | 440 | 465
Percentage of Participants | 0.2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.2 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Sequence 1: MK-0524B 1.8g/20mg vs Sequence 2: MK-0524A 2g+Simvastatin 20mg; Periods I/II; Test type: Superiority or Other; Difference in Percentage = 0.2, 95% CI 2-sided [-0.5 to 0.9] — Wilson's Score Method
Statistical Analysis 2: Comparison: Sequence 3: MK-0524B 1.8g/40mg vs Sequence 4: MK-0524A 2g+Simvastatin 40mg; Periods I/II; Test type: Superiority or Other; Difference in Percentage = -0.2, 95% CI 2-sided [-0.9 to 0.5] — Wilson's Score Method

16. Secondary Outcome: Percentage Change From Baseline in LDL-C at Week 4
Description: Blood samples taken at baseline (Day1 of Period I) and after 4 weeks of treatment to determine the LDL-C levels. The change from baseline after 4 weeks of treatment was recorded.
Time Frame: Baseline (Day1 of Period I) and Week 4
Population: Participants that completed the study and had respective endpoint data available at baseline and end of each treatment period. End of period value was defined as measurements collected on the same date as the corresponding end of period visit date. Results were reported by dose of study drug taken and not by randomly assigned sequence.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Groups:
- MK-0524B 0.9g/10mg: Participants who received MK-0524B 0.9g/10mg for 4 weeks in Period I regardless of randomly assigned sequence.
- MK-0524A 1g+Simvastatin 10mg: Participants who received MK-0524A 1g+Simvastatin 10mg for 4 weeks in Period I regardless of randomly assigned sequence.
- MK-0524B 0.9 g/40 mg: Participants who received MK-0524B 0.9g/40mg for 4 weeks in Period I regardless of randomly assigned sequence.
- MK-0524A 1 g + Simvastatin 40 mg: Participants who received MK-0524A 1g+Simvastatin 40mg for 4 weeks in Period I regardless of randomly assigned sequence.
Arm/Group | MK-0524B 0.9g/10mg | MK-0524A 1g+Simvastatin 10mg | MK-0524B 0.9 g/40 mg | MK-0524A 1 g + Simvastatin 40 mg
Number analyzed (Participants) | 582 | 574 | 556 | 581
Percentage Change | -34.8 [-36.6 to -33.0] | -35.8 [-37.6 to -34.0] | -42.2 [-44.3 to -40.0] | -45.8 [-48.0 to -43.7]
Statistical Analysis 1: Comparison: MK-0524B 0.9g/10mg vs MK-0524A 1g+Simvastatin 10mg; Test type: Superiority or Other; p = 0.341, ANOVA; Factors for treatment, country and gender; Difference in Least Squares Means = 1.0, 95% CI 2-sided [-1.1 to 3.1]
Statistical Analysis 2: Comparison: MK-0524B 0.9 g/40 mg vs MK-0524A 1 g + Simvastatin 40 mg; Test type: Superiority or Other; p = 0.004, ANOVA; Factors for treatment, country and gender; Difference in Least Squares Means = 3.7, 95% CI 2-sided [1.2 to 6.1]

17. Secondary Outcome: Percentage Change From Baseline in HDL-C at Week 4
Description: Blood samples taken at baseline (Day1 of Period I) and after 4 weeks of treatment to determine the HDL-C levels. The change from baseline after 4 weeks of treatment was recorded.
Time Frame: Baseline (Day1 of Period I) and Week 4
Population: as for outcome 16
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | MK-0524B 0.9g/10mg | MK-0524A 1g+Simvastatin 10mg | MK-0524B 0.9 g/40 mg | MK-0524A 1 g + Simvastatin 40 mg
Number analyzed (Participants) | 582 | 575 | 555 | 583
Percentage Change | 18.3 [16.6 to 19.9] | 18.7 [17.0 to 20.3] | 19.8 [17.9 to 21.6] | 19.6 [17.8 to 21.4]
Statistical Analysis 1: Comparison: MK-0524B 0.9g/10mg vs MK-0524A 1g+Simvastatin 10mg; Test type: Superiority or Other; p = 0.690, ANOVA; Factors for treatment, country and gender; Difference in Least Squares Mean = -0.4, 95% CI 2-sided [-2.3 to 1.5]
Statistical Analysis 2: Comparison: MK-0524B 0.9 g/40 mg vs MK-0524A 1 g + Simvastatin 40 mg; Test type: Superiority or Other; p = 0.879, ANOVA; Factors for treatment, country and gender; Difference in Least Squares Means = 0.2, 95% CI 2-sided [-1.9 to 2.3]

ADVERSE EVENTS:
Time Frame: up 20 weeks (12 weeks in Period I/II and 8 weeks in Period III)
Description: All participants who received at least 1 dose of study drug. Safety analysis was based on the experiences accumulated during Periods I/II combined (pre-crossover), where the study follows a parallel design. A separate safety analysis was performed for Period III (post-crossover).
Groups:
- Sequence 2: MK-0524A 2g+Simvastatin 20mg: Participants who received MK-0524B 1g + Simvastatin 20mg and MK-0524B 2g+ Simvastatin 20mg during Periods I/II
- Sequence 1: MK-0524A 2g+Simvastatin 20mg: Participants who received MK-0524B 1g + Simvastatin 20mg and MK-0524B 2g+ Simvastatin 20mg during Period III
Arm/Group | Sequence 1: MK-0524B 1.8g/20mg | Sequence 2: MK-0524A 2g+Simvastatin 20mg | Sequence 1: MK-0524A 2g+Simvastatin 20mg | Sequence 2: MK-0524B 1.8g/20mg | Sequence 3: MK-0524B 1.8g/40mg | Sequence 4: MK-0524A 2g+Simvastatin 40mg | Sequence 3: MK-0524A 2g+Simvastatin 40mg | Sequence 4: MK-0524B 1.8g/40mg
Serious Adverse Events (participants affected / at risk) | 3/610 | 6/602 | 4/472 | 2/440 | 12/597 | 9/605 | 4/440 | 3/465
Other Adverse Events (participants affected / at risk) | 225/610 | 227/602 | 40/472 | 48/440 | 222/597 | 237/605 | 31/440 | 45/465
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sequence 1: MK-0524B 1.8g/20mg (N=610) | Sequence 2: MK-0524A 2g+Simvastatin 20mg (N=602) | Sequence 1: MK-0524A 2g+Simvastatin 20mg (N=472) | Sequence 2: MK-0524B 1.8g/20mg (N=440) | Sequence 3: MK-0524B 1.8g/40mg (N=597) | Sequence 4: MK-0524A 2g+Simvastatin 40mg (N=605) | Sequence 3: MK-0524A 2g+Simvastatin 40mg (N=440) | Sequence 4: MK-0524B 1.8g/40mg (N=465)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device migration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sequence 1: MK-0524B 1.8g/20mg (N=610) | Sequence 2: MK-0524A 2g+Simvastatin 20mg (N=602) | Sequence 1: MK-0524A 2g+Simvastatin 20mg (N=472) | Sequence 2: MK-0524B 1.8g/20mg (N=440) | Sequence 3: MK-0524B 1.8g/40mg (N=597) | Sequence 4: MK-0524A 2g+Simvastatin 40mg (N=605) | Sequence 3: MK-0524A 2g+Simvastatin 40mg (N=440) | Sequence 4: MK-0524B 1.8g/40mg (N=465)
Diarrhoea (Gastrointestinal disorders) | 28 (32) | 33 (41) | 10 (10) | 15 (17) | 27 (29) | 37 (39) | 8 (8) | 13 (15)
Headache (Nervous system disorders) | 18 (19) | 32 (35) | 5 (6) | 9 (10) | 24 (25) | 28 (31) | 6 (8) | 8 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 67 (79) | 72 (84) | 9 (11) | 15 (17) | 50 (54) | 75 (93) | 5 (5) | 7 (7)
Flushing (Vascular disorders) | 155 (189) | 132 (166) | 23 (34) | 15 (20) | 162 (189) | 151 (179) | 14 (15) | 19 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.